CLINICAL TRIAL: NCT01853059
Title: Observational Study of Functional Outcomes After Chemoradiotherapy for Squamous Cell Cancer of the Anus
Brief Title: Functional Outcomes Following Anal Cancer Treatment
Acronym: FOFACT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: The Christie NHS Foundation Trust (Other); Bowel Disease Research Foundation (Unknown)
Responsible Party: Principal Investigator, Adam Stearns, Specialist Registrar in Surgery, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: A092896
Record Dates: First submitted 2013-05-10; First posted 2013-05-14 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Anal Cancer
Keywords: Anal cancer; Squamous cell cancer; Radiotherapy; Chemoradiotherapy; Conformational radiotherapy; Intensity modulated radiation therapy; IMRT
MeSH Terms: conditions — Anus Neoplasms; Neoplasms, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IMRT: Prospective longitudinal assessment of patients receiving intensity-modulated radiation therapy for anal cancer
- Conventional: Cross-sectional analysis of patients receiving conventional radiotherapy

SUMMARY:
Anal cancer is treated with chemoradiotherapy- combined chemotherapy and radiotherapy. This is very successful (75% long term survival). During the course of the radiotherapy, other organs in the pelvis may be damaged. This can lead to long-term problems with possible changes to the skin, bowels with diarrhoea and incontinence problems, bladder shrinkage and incontinence of urine, sexual problems including impotence and ejaculatory problems, or pain during sexual intercourse with vaginal dryness and shrinkage. Patients should be offered help with these side effects. At present, there is very little information on the effect treatment has on a patient's quality of life, making it difficult to judge if new treatment methods are better.

This project will measure quality of life from the patient's perspective after treatment for anal cancer. It will also gather preliminary data on quality of life after the introduction of a new technique for more precise 3D-targeting of radiotherapy beams at the cancer, called IMRT.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Squamous cell or basaloid carcinoma of the anal canal

Exclusion Criteria:

* adenocarcinoma, melanoma, lymphoma, sarcoma or other malignancy of anal canal
* Any synchronous or metanchronous pelvic malignancy of non-anal origin (eg. prostatic, genital tract)
* unable to complete questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under the care of the anal cancer multidisciplinary team in Addenbrookes, Cambridge and Christie Hospital, Manchester
Sampling Method: Non-Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Functional quality of life after chemoradiotherapy for anal cancer | 3 years
  Quality of life measured using:
  General
  * EORTC (European Organisation for Research and Treatment of Cancer) QLQ-C30
  Disease specific
  * EORTC QLQ-CR29
  * Vaizey incontinence score
  * MOS (Medical Outcomes Survey) sexual questionnaire

SECONDARY OUTCOMES:
Patient-reported treatment-related toxicity after chemoradiotherapy for anal cancer | 3 years
  Patient-reported treatment related toxicity measured with:
  * Common Terminology Criteria for Adverse Events (CTCAE version 3)
  * Pelvis questionnaire male & female (LENT/SOMA)
  (LENT/SOMA: see Barraclough LH et al. Radiother Oncol; 103:327-32)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Addenbrookes Hospital, Cambridge
  - Christie Hospital, Manchester

REFERENCES:
- [Background] Provencher S, Oehler C, Lavertu S, Jolicoeur M, Fortin B, Donath D. Quality of life and tumor control after short split-course chemoradiation for anal canal carcinoma. Radiat Oncol. 2010 May 23;5:41. doi: 10.1186/1748-717X-5-41. PMID 20492729
- [Background] Brown MW, Brooks JP, Albert PS, Poggi MM. An analysis of erectile function after intensity modulated radiation therapy for localized prostate carcinoma. Prostate Cancer Prostatic Dis. 2007;10(2):189-93. doi: 10.1038/sj.pcan.4500938. Epub 2006 Dec 26. PMID 17189954
- [Background] Barraclough LH, Routledge JA, Farnell DJ, Burns MP, Swindell R, Livsey JE, Davidson SE. Prospective analysis of patient-reported late toxicity following pelvic radiotherapy for gynaecological cancer. Radiother Oncol. 2012 Jun;103(3):327-32. doi: 10.1016/j.radonc.2012.04.018. Epub 2012 May 23. PMID 22633812